CLINICAL TRIAL: NCT00438828
Title: Dexamethasone for the Prophylaxis of Radiation-Induced Pain Flare Following Palliative Radiotherapy for Bone Metastases
Brief Title: Dexamethasone for the Prophylaxis of Pain Flare Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Edward Chow, Professor, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-14-0055; Sunnybrook REB# 057-2008 (Other: Sunnybrook Health Sciences Centre)
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Cancer
Keywords: radiation therapy; palliative; pain
MeSH Terms: conditions — Neoplasms; Pain | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexamethasone (Experimental): 8mg Dexamethasone PO on days 0 (prior to radiation treatment), and days 1, 2, and 3 following radiation treatment.
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — 8mg Dexamethasone PO on days 0 (prior to radiation treatment), and days 1, 2, and 3 following radiation treatment.
  Other Names: Decadron

SUMMARY:
Radiation treatment is often recommended as a safe and quick treatment that gives most people good relief from bone pain within a couple of weeks. However, some people can experience a short episode of increased pain (called a 'flare') a day or two after radiation treatment, that lasts about a day. The purpose of this sturdy is to find out if a medication called dexamethasone can help prevent pain flare as a result of radiation therapy.

DETAILED DESCRIPTION:
Of all people diagnosed with cancer, 25% will have their cancer come back and spread to the bones. This often results in significant pain and suffering. Radiation treatment is often recommended as a safe and quick treatment that gives most people good relief from bone pain within a couple of weeks. However, some people can experience a short episode of increased pain called a flare a day or two after radiation treatment that lasts about a day. Studies suggest that around a third of all people who receive radiation treatment to help pain from cancer in the bones will have a pain flare. This study is being done because it would be helpful to prevent extra bone pain from happening to people after they receive radiation treatments. The purpose of this study is to find out if a medication called dexamethasone can help prevent pain flare as a result of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented bone metastases by radiological imaging
* Patients at least 18 years of age
* Written consent
* KPS ≥ 40
* Baseline worst pain at the planned radiated bony metastatic site ≥ 2
* Patient able to inform the pain score at the planned radiated bony metastatic site

Exclusion Criteria:

* Concurrent use of any corticosteroid medication other than topical or inhaled preparations
* Medical contraindications to corticosteroids such as diabetes mellitus, uncontrolled hypertension or active peptic ulcer
* Pathological fracture of the irradiated extremity
* Spinal cord compression
* Language barrier
* Immediate change in regular analgesic medication. If the oncologist thinks the patient is not receiving adequate analgesic, we recommend the oncologist to increase the analgesic first to stabilize ot lessen the pain before recruiting the patient to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Complete control of pain flare on days 1-5 after the completion of radiation treatment. | Days 1-5

SECONDARY OUTCOMES:
Complete control of pain flare from Day 6-10 after the completion of radiation treatment. | Days 6-10
Functional interference especially mood and sleep in Brief Pain Inventory will be monitored. | Days 0, 1-10, and 6-weeks from baseline assessment
Quality of life outcomes | Baseline and 6-weeks following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chow, MBBS PhD, Study Chair — edward.chow@sunnybrook.ca
Locations (1):
- Odette Cancer Centre, Toronto, Ontario, Canada